CLINICAL TRIAL: NCT05477875
Title: Randomized, Controlled Cross-over Comparison of Cannabinoid to Oral Opioid for Postoperative Photorefractive Keratectomy Pain Control
Brief Title: Cannabinoid vs Opioid for Photorefractive Keratectomy Pain Control
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Consortium for Medical Marijuana Clinical Outcomes Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB202201660 -A
Record Dates: First submitted 2022-07-21; First posted 2022-07-28 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-06

CONDITIONS: Photorefractive Keratectomy; Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia | interventions — Cannabinoids; Dronabinol; acetaminophen, codeine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral cannabinoid (Experimental): Oral cannabinoid
  Interventions: Drug: oral cannabinoid
- Oral codeine/acetaminophen (Active Comparator): Oral codeine-acetaminophen for controlling pain
  Interventions: Combination Product: oral codeine/acetaminophen

INTERVENTIONS:
Drug: oral cannabinoid — dronabinol
  Other Names: dronabinol
  Arms: Oral cannabinoid
Combination Product: oral codeine/acetaminophen — 10 tablets of acetaminophen-codeine combination (300-30mg) without refills.
  Arms: Oral codeine/acetaminophen

SUMMARY:
Photorefractive Keratectomy (PRK) is a commonly performed corneal refractive surgery but has significant post-operative pain. Pain medications after PRK are typically opioid-acetaminophen combinations. Alternatives to opioid medication are worth consideration. Patients will receive PRK in each eye sequentially, using the cannabinoid or codeine/acetaminophen for one eye and the other treatment for the fellow eye two weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 18 years with refractive stability for 1 year electing to have PRK surgery
* Consenting to participate
* Not meeting exclusion criteria will be included in the study population.

Exclusion Criteria:

* Patients not candidates for PRK will be excluded from the study.
* Patients taking other pain medications for concomitant medical conditions including, but not limited to tricyclic antidepressants, gabapentin and tramadol will be excluded from the study.
* Additional exclusion criteria will be known or suspected allergy or hypersensitivity to any of the routine or study medications.
* Patients completing follow up appointments at anywhere other than UF Health Ophthalmology clinic at the Oaks will not be enrolled in the study.
* Patients who are pregnant or nursing are not eligible for PRK, and such patients are not eligible to enroll in this study. Female patients of child-bearing age will be pregnancy tested before surgery and study enrollment.
* Patients will be specifically counseled, and it will be noted in the written informed consent that use of the cannabinoid product may result in a positive THC urinalysis screening test so they may self-exclude if such a situation could cause social and/or employment conflict.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W Steigleman, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Oaks Eye Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-five myopic patients were recruited and had surgery for both eyes completed between 1/1/2024 and 12/31/2024. Patients seeking refractive surgery and who were candidates for photorefractive keratectomy were approached with the option to enroll in the ophthalmology clinic.
Pre-assignment Details: Any patient who could not undergo surgery due to contraindications such as thin cornea, irregular astigmatism, or inability to lay flat were excluded. Patients who could not undergo sequential eye surgery due to scheduling constraints could not enroll in the study.
Groups:
- Group 1: Group 1 patients were assigned to take CBD 50mg 2x/day by mouth for 1 week after surgery on the first eye and Tylenol T3 30-300mg 3x/day by mouth for 1 week after surgery on the fellow eye.
- Group 2: Group 2 patients were assigned to take Tylenol T3 30-300mg 3x/day by mouth for 1 week after surgery on the first eye and CBD 50mg 2x/day by mouth for 1 week after surgery on the fellow eye.
Period: Preoperative
Arm/Group | Group 1 | Group 2
Started | 16 | 19
Completed | 16 | 19
Not Completed | 0 | 0
Period: POW1
Arm/Group | Group 1 | Group 2
Started | 16 | 19
Completed | 16 | 19
Not Completed | 0 | 0
Period: POM1
Arm/Group | Group 1 | Group 2
Started | 16 | 19
Completed | 16 | 19
Not Completed | 0 | 0
Period: POM3
Arm/Group | Group 1 | Group 2
Started | 16 | 19
Completed | 16 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Group 1 patients had 50mg CBD chemovar twice a day by mouth after their first photorefractive surgery on one eye, then later had Tylenol T3 30-300mg three times a day by mouth after their second surgery on the fellow eye.
- Group 2: Group 2 patients had Tylenol T3 30-300mg three times a day by mouth after their first photorefractive surgery on one eye, then later had 50mg CBD chemovar twice a day by mouth after their second surgery on the fellow eye.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] — Because patients were their own controls, age is unchanged across groups.
  Years | 34.2 (5.2) | 30.6 (6.8) | 32.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Because patients were their own controls, demographics are unchanged across groups.
  Participants
    Female | 9 | 10 | 19
    Male | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants] — Not recorded.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 16 | 19 | 35
Visual Acuity [Mean (Standard Deviation); unit: LogMAR] — Vision measured for the eye operated on under each drug. Population: Crossover study, so participants were their own controls.
  LogMAR
    without glasses or contacts | 1.109 (0.452) | 1.290 (0.475) | 1.207 (0.470)
    With glasses or contacts | -0.062 (0.085) | 0.026 (0.338) | -0.014 (0.257)

OUTCOME MEASURES:

1. Primary Outcome: Pain as Recorded by the FACES Scale (Maximum) After First Surgery
Description: The Wong-Baker Faces Pain Rating Scale is a pain scale that was developed by Donna Wong and Connie Baker. The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable"
Time Frame: 1 week after first surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cannabidiol: Patients given 50mg CBD chemovar twice a day by mouth after photorefractive surgery on one eye. Depending on study group, this may be after the first or second surgery.
- Tylenol T3: Patients given Tylenol T3 30-300mg three times a day by mouth after photorefractive surgery on one eye. Depending on study group, this may be after the first or second surgery.
Arm/Group | Cannabidiol | Tylenol T3
Number analyzed (Participants) | 16 | 19
units on a scale | 1.33 (0.95) | 1.27 (0.89)
Statistical Analysis 1: Comparison: Cannabidiol vs Tylenol T3; Test type: Equivalence — Two-way ANOVA using group and intervention as fixed factors were analyzed, with outcome variable p-value reported below, threshold 0.05; p = 0.538, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Pain as Recorded by the FACES Scale (Maximum) After Second Surgery
Description: as for outcome 1
Time Frame: 1 week after second surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cannabidiol | Tylenol T3
Number analyzed (Participants) | 19 | 16
units on a scale | 1.46 (0.82) | 1.79 (1.12)
Statistical Analysis 1: Comparison: Cannabidiol vs Tylenol T3; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.538, ANOVA

3. Secondary Outcome: Uncorrected Visual Acuity of First Eye Surgery
Description: Uncorrected visual acuity as measured by Snellen Chart
Time Frame: 3 months after first surgery
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Cannabidiol | Tylenol T3
Number analyzed (Participants) | 16 | 19
LogMAR | -0.123 (0.119) | -0.054 (0.169)
Statistical Analysis 1: Comparison: Cannabidiol vs Tylenol T3; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.516, ANOVA

4. Secondary Outcome: PROWL-SS
Description: An online questionnaire derived from the Patient-Reported Outcomes With LASIK (PROWL) will be given to patients after PRK at 3 months. It ranges from 0-100, where 100 indicates best possible vision and satisfaction, while 0 indicates worst possible vision and satisfaction.
Time Frame: 3 month
Population: Surveys assess overall quality of life which cannot be specifically attributed to a single eye since vision is binocular. For example, having excellent vision in one eye and poor vision in the other can be more disturbing than having poor vision in both eyes or cause patients to suffer from double vision. Because all survey measurements are implied to be binocular at 3 months after both surgeries are done, results are displayed by group instead of intervention. There is no separate measurement.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 16 | 19
score on a scale
  Pre-op | 58.0 (20.1) | 60.9 (18.3)
  Post-op Month 3 | 81.6 (9.0) | 85.6 (6.9)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Equivalence — Alpha = 0.05, two-way ANOVA with "Group" x "Time Points" as fixed factors and PROWL-SS from (1-100) as the dependent variable; p < 0.851, ANOVA

5. Secondary Outcome: Quality of Life Refractive Correction Survey
Description: The QIRC measures quality of life associated with vision and eyewear problems, measured at 3 months. It ranges from 0-100, where 0 indicates best possible vision and quality of life and 100 indicates worst possible vision and quality of life.
Time Frame: 3 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 16 | 19
score on a scale
  Pre-op | 37.7 (6.2) | 37.6 (10.6)
  Post-op Month 3 | 19.2 (6.0) | 26.4 (6.3)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Equivalence — Alpha = 0.05, two-way ANOVA with "Group" x "Time Points" as fixed factors and QIRC from (1-100) as the dependent variable; p < 0.543, ANOVA

6. Secondary Outcome: Ocular Discomfort Questionnaire
Description: An online questionnaire derived from the Ocular Surface Disease Index (OSDI) at 3 months. It ranges from 0-48, where 0 indicates no eye discomfort and 48 indicates constant, debilitating, worst-possible eye discomfort or pain.
Time Frame: 3 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 16 | 19
score on a scale
  Pre-op | 4.9 (5.7) | 4.8 (5.4)
  Post-op Month 3 | 4.9 (4.8) | 3.9 (4.0)
Statistical Analysis 1: Comparison: Group 1; Test type: Equivalence — Alpha = 0.05, two-way ANOVA with "Group" x "Time Points" as fixed factors and OSDI from (0-48) as the dependent variable; p = 0.725, ANOVA

7. Secondary Outcome: Uncorrected Visual Acuity of Second Eye Surgery
Description: Uncorrected visual acuity as measured by Snellen Chart
Time Frame: 3 months after second surgery
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Cannabidiol | Tylenol T3
Number analyzed (Participants) | 19 | 16
LogMAR | -0.051 (0.16) | -0.075 (0.121)
Statistical Analysis 1: Comparison: Cannabidiol vs Tylenol T3; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.516, ANOVA

ADVERSE EVENTS:
Time Frame: 3 months
Description: Patients are not expected to die from photorefractive keratectomy nor are serious adverse events generally expected.
Arm/Group | Cannabidiol | Tylenol T3
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

LIMITATIONS AND CAVEATS:
This study could not separate the effects of long-term vision quality of life outcomes between drugs, although these secondary outcomes are only for safety monitoring and not for comparing drug effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT05477875/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT05477875/SAP_001.pdf
  • Informed Consent Form (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT05477875/ICF_002.pdf